CLINICAL TRIAL: NCT04708847
Title: A Double-Blind, Placebo-Controlled, Randomized Clinical Pharmacology Study to Evaluate the Prevention Effect and the Recovery-Promoting Effect of a Single Subcutaneous Administration of GYM329 on Disuse Muscle Atrophy in Healthy Male Volunteers
Brief Title: A Clinical Pharmacology Study to Evaluate the Effect of GYM329 on Disuse Muscle Atrophy in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JP42791
Record Dates: First submitted 2020-12-24; First posted 2021-01-14 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pre-immobilization active drug group (Experimental): Subjects will receive a single subcutaneous dose of GYM329 on Day 1 and a single subcutaneous dose of placebo on Day 15.
  Interventions: Drug: GYM329
- Post-immobilization active drug group (Experimental): Subjects will receive a single subcutaneous dose of placebo on Day 1 and a single subcutaneous dose of GYM329 on Day 15.
  Interventions: Drug: GYM329
- Placebo group (Placebo Comparator): Subjects will receive a single subcutaneous dose of placebo on Day 1 and a single subcutaneous dose of placebo on Day 15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GYM329 — GYM329 subcutaneous injection
  Arms: Post-immobilization active drug group; Pre-immobilization active drug group
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo group

SUMMARY:
This study will induce disuse atrophy through unilateral immobilization of the thigh and lower leg in healthy male volunteers to evaluate the PD of a single subcutaneous dose of GYM329 prior to or after unilateral thigh and lower leg immobilization.

Healthy male volunteers will receive either GYM329 or placebo by subcutaneous injection at two time points, before and after 2 weeks of unilateral thigh and lower leg immobilization, in an investigator- and subject-blinded, randomized, placebo-controlled, parallel-group design. At enrollment, all subjects will be randomized in a 1:2 ratio to either the pre-immobilization active drug group receiving a single subcutaneous dose of GYM329 before unilateral thigh and lower leg immobilization (Group A) or the pre-immobilization placebo group receiving a single subcutaneous dose of placebo before unilateral thigh and lower leg immobilization (Group B). On Day 15, subjects assigned to Group B and who completed the muscle strength assessment at Day15 will be further randomized in a 1:1 ratio to either the post-immobilization active drug group (Group B-1) or the post-immobilization placebo group (Group B-2). Group A will receive GYM329 on Day 1 and placebo on Day 15. Group B will receive placebo on Day 1. Subsequently, Group B-1 will receive GYM329 on Day 15 and Group B-2 will receive placebo on Day 15.

Muscle strength will be measured at pre-immobilization of unilateral thigh and lower leg, post-immobilization of unilateral thigh and lower leg (Day 15), Day 29, and Day 43. Subjects will be observed for 252 days after the second study treatment administration (266 days after the first study treatment administration).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and to comply with the study protocol
* Healthy men aged from 18 to less than 40 years at the time of consent
* Right leg dominant
* Agreed to limit physical activity as directed by study site staff from the time of informed consent until the end of the muscle strength evaluation period (completion of Day 43)
* BMI is between 18.5 and less than 25.0 at screening
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.

Exclusion Criteria:

* History of congenital myopathy
* Congenital thrombophilia
* Previous or current VTE
* History of hip or limb surgery, spine or spinal cord surgery, or laparotomy (excluding laparotomy for appendicitis or inguinal hernia), or laparoscopic surgery (e.g. cholecystectomy)
* History of fracture of the pelvis or open/compound fracture of lower limb, or history of fracture within 3 years prior to screening, excluding digit fracture
* History of severe trauma, trauma requiring surgical intervention, or trauma with organ injury which deemed as clinically significant by the investigator
* Previous or current medical condition that could lead to thrombosis as judged by the investigator
* Angiography within 6 months before first study treatment administration
* Current Grade ≥ 3 thermal burn or history of Grade ≥ 3 thermal burn within 3 months prior to study treatment administration
* Unable to wear compression stockings
* History of heparin-induced thrombocytopenia or hypersensitivity to the LMWH and to the heparin or any other clinically significant contra-indications for use of LMWH
* Participation in bodybuilding or full time employment in a physically demanding occupation
* Immobilization, surgery, or traumatic injury of the arm within 90 days before first study treatment administration
* Traumatic injury of the leg within 6 months before first study treatment administration
* Immobilization or surgery of the leg within 6 months before first study treatment administration
* Immobilization of the leg for 2 or more weeks within 12 months before first study treatment administration
* Contraindication for MRI
* Habitual excessive over- or under-eating
* Any condition that may interfere with assessment of local pain and pruritus at the injection site

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Thigh muscle strength score | 28 days
  Percent change in thigh muscle strength score from Day 1 to Day 15 and Day 15 to Day 29 (Thigh muscle strength score: peak isometric knee extension torque and peak isokinetic knee extension torque at 90°/s and 180°/s)

SECONDARY OUTCOMES:
Safety; Adverse event monitoring | 45 weeks
  Incidence and severity of adverse events
Safety; Laboratory tests | 45 weeks
  Incidence of laboratory abnormalities, based on clinical laboratory tests
Safety; Vital signs | 45 weeks
  Abnormality in vital signs
Safety; Electrocardiogram (ECG) | 45 weeks
  Abnormality in Electrocardiograms (ECGs)
Pharmacokinetics; Serum GYM329 concentrations | 45 weeks
  Serum GYM329 concentrations over time
Pharmacokinetics; Cmax | 45 weeks
  Cmax of GYM329
Pharmacokinetics; Tmax | 45 weeks
  Tmax of GYM329
Pharmacokinetics; AUC | 45 weeks
  AUC of GYM329
Pharmacokinetics; T1/2 | 45 weeks
  T1/2 of GYM329
Immunogenicity | 45 weeks
  Incidence of serum anti-GYM329 antibodies
Pharmacodynamics; Muscle volume | 45 weeks
  Changes in thigh muscle volume over time
Pharmacodynamics; Total and free latent myostatin, mature myostatin | 45 weeks
  Changes in total and free latent myostatin, mature myostatin over time

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).